CLINICAL TRIAL: NCT02425072
Title: NovoTTFTM-100A System Therapy for Refractory CNS Involved Small Cell Lung Cancer
Brief Title: NovoTTF-100A Therapy for Refractory CNS Involved Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: John Villano (Other)
Responsible Party: Sponsor-Investigator, John Villano, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-NEURO-05-MCC
Record Dates: First submitted 2014-12-11; First posted 2015-04-23 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Small Cell Lung Cancer; Brain Metastasis
Keywords: Cancer; Brain; Lung; Small-cell
MeSH Terms: conditions — Small Cell Lung Carcinoma; Brain Neoplasms; Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NovoTTF-100A plus chemotherapy (Experimental): NovoTTF-100A System with Physician's Choice Chemotherapy
  Interventions: Device: NovoTTF-100A plus chemotherapy

INTERVENTIONS:
Device: NovoTTF-100A plus chemotherapy — NovoTTF-100A System with Physician's Choice Chemotherapy

SUMMARY:
The hypothesis of this study is that the addition of NovoTTF-100A System treatment to salvage chemotherapy will significantly increase time to treatment failure in the brain of small cell lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed small cell lung cancer histology with CNS metastases
* Parenchymal disease, ten or less lesions, and supratentorial
* PS 70% or greater
* Prior CNS radiotherapy.
* No previous or currently active second malignancy
* Age > 22 years.
* Life expectancy of ≥ 3 months.

Exclusion Criteria:

* Significant liver function impairment - AST or ALT > 3 times the upper limit of normal; Total bilirubin > upper limit of normal.
* Significant renal impairment (serum creatinine > 1.7 mg/dL).
* Coagulopathy (as evidenced by PT or APTT >1.5 times in control patients not undergoing anticoagulation).Thrombocytopenia (platelet count < 100 x 103/μL).
* Neutropenia (absolute neutrophil count < 1 x 103/μL).
* Anemia (Hb < 10 g/L).
* Severe acute infection. Serious non-healing wound or ulcer on scalp
* Significant co-morbidities within 4 weeks prior to enrollment.
* Implanted pacemaker, defibrillator or deep brain stimulator, or documented clinically significant arrhythmias.
* Active implanted medical device (e.g. deep brain stimulators, spinal cord stimulators, vagus nerve stimulators, pacemakers, defibrillators, and programmable shunts).
* Skull defect (e.g. missing bone with no replacement).
* Shunt
* Bullet fragments
* Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness).
* Sensitivity to conductive hydrogels.
* Pregnant or lactating women

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure | Up to 3 months

SECONDARY OUTCOMES:
Progression Free Survival | Up to 6 months
Overall response rate | Up to 2 years
Duration of response | Up to 2 years
Safety of treatment assessed by number of participants with adverse events | Up to 2 years
  As a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: John L Villano, MD, PhD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky, Markey Cancer Center, Lexington, Kentucky, United States